CLINICAL TRIAL: NCT06596772
Title: A Prospective, Randomized, Double-blind, Parallel-group Study to Compare the Efficacy, Safety, Pharmacokinetics and Immunogenicity of MB04 and EU-sourced Enbrel® in Patients with Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study to Compare Efficacy, Pharmacokinetics, Safety and Immunogenicity of MB04 [proposed Etanercept Biosimilar] to Enbrel® [EU-sourced] in Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB04-C-01-23
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MB04 (proposed etanercept biosimilar) (Experimental): MB04 50 mg/week via subcutaneous injection
  Interventions: Drug: MB04 (proposed biosimilar to etanercept)
- Enbrel (etanercept) (Active Comparator): Enbrel 50 mg/week via subcutaneous injection
  Interventions: Drug: Enbrel (etanercept)

INTERVENTIONS:
Drug: MB04 (proposed biosimilar to etanercept) — MB04 50 mg/week via subcutaneous injection
  Arms: MB04 (proposed etanercept biosimilar)
Drug: Enbrel (etanercept) — Enbrel 50 mg/week via subcutaneous injection
  Arms: Enbrel (etanercept)

SUMMARY:
A study to compare efficacy, pharmacokinetics, safety and immunogenicity of MB04 [proposed etanercept biosimilar] to Enbrel® [EU-sourced] in rheumatoid arthritis

DETAILED DESCRIPTION:
The study will randomize approximately 458 patients aged between 18 and 75 years with active Rheumatoid Arthritis despite methotrexate therapy.

All patients shall receive methotrexate for ≥12 weeks and on a stable dose (10 to 25 mg/week) for ≥8 weeks prior to randomization, and folic acid (≥5 mg/week) from 4 weeks prior to screening until the end of the treatment period (Week 36).

Screening evaluations will be completed within 28 days prior to randomization. There will be 2 periods in the study: Main Treatment period and Transition period.

During the Main Treatment Period, eligible patients will be randomized, at a 1:1 ratio, to administer a 50 mg weekly dose of MB04 or EU- sourced Enbrel® subcutaneously (SC) using an Interactive Response System (IRT). After completing Week 24 assessment, patients will continue to receive the study treatment up to Week 36. Those patients who were originally assigned to EU-sourced Enbrel® will be randomized, at a 1:1 ratio, to receive either MB04 or EU-sourced Enbrel® SC, while patients originally assigned to MB04 will continue with the same treatment until Week 36.

After treatment discontinuation, patients will undergo a Safety follow-up period for 4 weeks, up to week 40.

ELIGIBILITY:
Inclusion

* Documented history of RA diagnosis consistent with the 2010 ACR/EULAR classification criteria ≥6 months prior to randomization (but not exceeding 15 years prior to screening).
* Moderately to severe RA despite appropriate MTX at baseline therapy defined as having more than or equal to six swollen joints and more than or equal to six tender joints and either erythrocyte sedimentation rate (ESR, Westergren) ≥ 28 mm/h or serum C-reactive protein > 5.0 mg/dL and positive rheumatoid factor and/or CCP at screening
* Stable dose MTX between 10 to 25 mg weekly during ≥12 weeks, since ≥8 weeks prior to randomization
* Stable dose of NSAID and /or other analgesics for at least 4 weeks prior to randomization, when used
* Stable dose ≤10 mg prednisone daily or equivalent for ≥4 weeks prior to randomization, when used
* Patients who are otherwise medically stable according to investigator's discretion
* Agree to use highly effective contraceptive methods up to 6 months after las dose Exclusion
* Previously treated with any biologic or targeted synthetic DMARD
* Previously treated with any monoclonal antibody for other condition than RA
* Hypersensitivity to any component of study drug and/or prefilled syringe components
* Arthritis with onset prior to age 16 years or current diagnosis of inflammatory joint disease other than RA
* Systemic manifestations of RA other that rheumatoid nodules or secondary Sjogren's syndrome
* Active infection or potentially relapsing infections that could have a severe outcome. Latent tuberculosis infection detected during screening should start an approved treatment regimen according to standard of care and rescreened
* Solid or hematologic malignancy within the past 5 years
* Pregnant and breastfeeding women
* Any medical condition in the opinion of the investigator that would be a risk for safety, cooperation in the study or interferes with the interpretation of the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
American College of Rheumatology 20% Response Criteria (ACR20) | Week 24

SECONDARY OUTCOMES:
ACR20 | Weeks 36
American College of Rheumatology 50% Response Criteria (ACR50) | Weeks 24 and 36
American College of Rheumatology 70% Response Criteria (ACR70) | Weeks 24 and 36

CONTACTS AND LOCATIONS:
Locations (60):
- Bulgaria (8):
  - Research site 2007, Haskovo
  - Research site 2005, Plovdiv
  - Research Site 2002, Rousse
  - Research site 2001, Sofia
  - Research Site 2003, Sofia
  - Research Site 2008, Sofia
  - Research site 2004, Vidin
  - Research site 2006, Vratsa
- Georgia (9):
  - Research site 7004, Batumi
  - Research site 7010, Batumi
  - Research site 7001, Tbilisi
  - Research site 7002, Tbilisi
  - Research site 7003, Tbilisi
  - Research site 7005, Tbilisi
  - Research site 7006, Tbilisi
  - Research site 7007, Tbilisi
  - Research site 7009, Tbilisi
- Moldova (2):
  - Research Site 1301, Chisinau
  - Research site 1302, Chisinau
- Poland (29):
  - Research Site 1603, Bialystok
  - Research Site 1614, Bialystok
  - Research site 1616, Bialystok
  - Research site 1613, Bydgoszcz
  - Research site 1623, Bytom
  - Research Site 1615, Elblag
  - Research Site 1627, Elblag
  - Research Site 1606, Gdynia
  - Research Site 1611, Katowice
  - Research Site 1617, Krakow
  - Research Site 1622, Lublin
  - Research site 1605, Nowa Sól
  - Research Site 1618, Opole
  - Research site 1628, Piotrkow Trybunalski
  - Research Site 1624, Poniatowa
  - Resarch Site 1619, Poznan
  - Research Site 1601, Poznan
  - Research Site 1602, Poznan
  - Research Site 1608, Poznan
  - Research Site 1621, Poznan
  - Research Site 1612, Siedlce
  - Research Site 1610, Sochaczew
  - Research site 1629, Stalowa Wola
  - Research Site 1620, Torun
  - Research Site 1604, Warsaw
  - Research Site 1607, Warsaw
  - Research Site 1609, Warsaw
  - Research Site 1625, Wroclaw
  - Research Site 1626, Zamość
- Romania (7):
  - Research Site 1803, Bacau
  - Research Site 1805, Brasov
  - Resarch Site 1801, Bucharest
  - Research site 1802, Bucharest
  - Research site 1804, Bucharest
  - Research site 1303, Chisináu
  - Research site 1806, Râmnicu Vâlcea
- Serbia (5):
  - Research site 1903, Belgrade
  - Research site 1904, Belgrade
  - Research site 1905, Belgrade
  - Research Site 1902, Novi Sad
  - Research site 1901, Zrenjanin

IPD SHARING:
Plan to Share IPD: Undecided